CLINICAL TRIAL: NCT06779500
Title: Pre-hospital Care in Burn Patients Presenting to Tertiary Care Centers of Nepal
Status: Completed | Type: Observational
Sponsor: Tribhuvan University Teaching Hospital, Institute Of Medicine. (Other)
Responsible Party: Principal Investigator, Ishwor Thapaliya, Mr., Tribhuvan University Teaching Hospital, Institute Of Medicine.
Other Study IDs: 2021-028
Record Dates: First submitted 2025-01-11; First posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Burns
Keywords: Burn injuries; Burn resuscitation; Pre-hospital care
MeSH Terms: conditions — Burns

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This cross-sectional study investigates pre-hospital practices among burn patients presenting to a tertiary care center in Nepal. It examines first aid measures, timelines to medical care, resuscitation protocols, and factors contributing to delays. Findings aim to highlight gaps in burn care and inform strategies to improve patient outcomes and management practices in resource-limited settings.

DETAILED DESCRIPTION:
Burn injuries are a major public health concern in low- and middle-income countries, contributing significantly to morbidity and disability-adjusted life years (DALYs) lost. This study focuses on understanding the pre-hospital care practices among burn patients in Nepal, a region with limited burn care resources and high incidence rates. Using structured interviews and clinical data, the study explores the type and adequacy of first aid provided, factors influencing delays in accessing tertiary care, and the effectiveness of initial resuscitation. By identifying gaps in awareness, infrastructure, and healthcare delivery, the study seeks to propose actionable recommendations for enhancing burn care systems and improving outcomes for burn patients in Nepal.

ELIGIBILITY:
Inclusion Criteria:

* Patients of all ages, genders, and backgrounds admitted to the study site with a primary diagnosis of burn injuries.

Exclusion Criteria:

* Patients with life-threatening injuries accompanying burns.
* Patients with a documented history of prior burn injuries.
* Individuals who decline to provide informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Burn patients presenting to a tertiary care center with diverse demographics, including variations in age, gender, socioeconomic status, and location, primarily from urban and rural settings in Nepal.
Sampling Method: Non-Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2021-11-12 (Actual); Primary Completion 2022-05-11 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Documentation of First Aid Practices Among Burn Patients | within 1st hour of burn
  This outcome evaluates the initial first aid measures applied by burn patients or their caregivers before reaching a tertiary care center, including the type, adequacy, and timing of interventions.

SECONDARY OUTCOMES:
Resuscitation Received in the First 24 Hours | First 24 hours after injury.
  Assesses the type, volume, and adequacy of resuscitation fluids administered within the initial 24-hour period following the burn injury.

CONTACTS AND LOCATIONS:
Locations (1):
- Ishwor Thapaliya, Kathmandu, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: Yes
The Individual Participant Data (IPD) from this study will be shared with other researchers upon reasonable request. Data to be shared will include de-identified participant data relevant to the study outcomes, including demographic information, first aid practices, treatment details, and timelines of burn care.
Supporting Information: Study Protocol
Time Frame: The data will be available beginning six months after publication and will remain accessible for three years.
Access Criteria: Researchers must submit a formal request, including a detailed research proposal and objectives, to the corresponding author. The request will be reviewed by the study team for approval. Data will be provided under a data-sharing agreement ensuring appropriate use and confidentiality.